CLINICAL TRIAL: NCT00138736
Title: Phase II Study on Mannan Binding Lectin (MBL) Substitution in MBL-Deficient Children With Chemotherapy-Induced Neutropenia
Brief Title: Study on Mannan Binding Lectin (MBL) Substitution in MBL-Deficient Children With Chemotherapy-Induced Neutropenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Collaborators: Landsteiner Foundation for Blood Transfusion (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KB2003.02
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2007-08

CONDITIONS: MBL-Deficient; Neutropenia
Keywords: MBL-deficient; chemotherapy; neutropenia; chemotherapy-induced neutropenia
MeSH Terms: conditions — Neutropenia | interventions — Mannose-Binding Lectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): MBL until the patient's absolute neutrophil count (ANC) is above 500/microL blood.
  Interventions: Drug: Mannan Binding Lectin (MBL); Drug: Mannan Binding Lectin

INTERVENTIONS:
Drug: Mannan Binding Lectin (MBL)
Drug: Mannan Binding Lectin — MBL dose at a twice weekly dose interval (3 or 4 days):
  0.2 mg/kg, for a 3-day interval; 0.3 mg/kg, for a 4-day interval
  Other Names: MBL SSI

SUMMARY:
The pharmacokinetics, and clinical and biological effects of MBL replacement therapy in MBL-deficient children during chemotherapy-induced neutropenia were studied.

DETAILED DESCRIPTION:
Mannan Binding Lectin (MBL) is a member of the lectin pathway of the complement system and plays an important role in the innate immune system. MBL replacement in MBL-deficient children with chemotherapy-induced neutropenia represents a new approach to lower the risk of febrile episodes, of hospital admission, of prolonged use of intravenous antibiotics and of severe infections.

The aim of the Phase II study is to find evidence for the correct prediction of plasma levels of MBL necessary for clinical effects and biological efficacy, to confirm the dosage regimen needed to reach the required MBL plasma levels, and reconfirm the safety and lack of side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 0 - 12 years, during chemotherapy, and expected to become neutropenic
* MBL deficiency by genotype or phenotype (< 100 ng/ml)
* Informed consent and assent of patient and/or legal representative

Exclusion Criteria:

* Inability or unwillingness to comply with the protocol or likely inability to complete the study period
* Known allergic reactions to MBL and other human plasma products
* Participation in other investigational drug studies within the last month
* Clinically relevant abnormalities in: serum immunoglobulins IgG, IgA, IgM; blood counts; complement factors measured by AP50, CH50; urine protein and cell counts; serum creatinine and liver enzymes, as routinely determined for regular patient care.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2004-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics of MBL | until the patient's absolute neutrophil count (ANC) is above 500/uL blood.

SECONDARY OUTCOMES:
days of fever | until the patient's absolute neutrophil count (ANC) is above 500/uL blood.
days of hospital admission | until the patient's absolute neutrophil count (ANC) is above 500/uL blood.
use of antibiotics or antifungal medication | until the patient's absolute neutrophil count (ANC) is above 500/uL blood.
number and type of infections | until the patient's absolute neutrophil count (ANC) is above 500/uL blood.
MBL-dependent opsonizing capacity in vitro | until the patient's absolute neutrophil count (ANC) is above 500/uL blood.
safety and incidence of side effects | until the patient's absolute neutrophil count (ANC) is above 500/uL blood.

CONTACTS AND LOCATIONS:
Overall Officials: T W Kuijpers, MD, PdD, Principal Investigator — Dept. of Paediatric Immunology, AMC, Amsterdam, The Netherlands; H N Caron, Principal Investigator — Dept of Paediatric Oncology, AMC, Amsterdam, The Netherlands
Locations (2):
- Netherlands (2):
  - Academic Medical Centre, Amsterdam
  - Erasmus Medical Centre, Rotterdam